CLINICAL TRIAL: NCT05557175
Title: A Mixed-methods Evaluation of the Clinical and Cost-effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) on Neurogenic Overactive Bladder in Stroke
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) on Neurogenic Overactive Bladder in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ref No. ZVSV
Record Dates: First submitted 2022-09-25; First posted 2022-09-27 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2022-09

CONDITIONS: Urgency Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Active and Sham rTMS groups
Who Masked: Participant, Care Provider
Masking Description: The therapist and the participants will be blinded in the recruitment, randomization and treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active rTMS group (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham rTMS group (Sham Comparator)
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — The active rTMS group will receive a 1 Hz inhibitory low-frequency rTMS protocol hotspot of the contra-lessional primary motor cortex (M1), will deliver a continuous pulse of 1 pulse per second totalling 1200 pulses of 80% active motor threshold stimulation. The duration of the stimulation will last for 20 minutes thrice a week for four weeks (12 sessions). The motor threshold will be the minimum single-pulse TMS intensity necessary to elicit a motor-evoked potential greater than 50μV in more than 5 out of 10 consecutive trials. The standard 70 mm figure-of-eight air-cooled coil handle (MagPro) will be held at right angle to the skull for effective M1 stimulation. The participants in the active rTMS groups will receive a subthreshold stimulation intensity for muscle contraction with no painful peripheral sensation
  Arms: Active rTMS group
Device: Sham rTMS — The sham rTMS will be applied using the same parameters as the active rTMS but the coil will be rotated 90° away from the scalp so that minimal or no flow of current will be induced
  Arms: Sham rTMS group

SUMMARY:
Neurogenic overactive bladder (NOAB) presents with urgency incontinence. Existing NOAB management is expensive, lacks standardized regimens, or is invasive. Therefore, evaluating the effectiveness of non-invasive repetitive transcranial magnetic stimulation (rTMS) for NOAB management among stroke survivors remains crucial.

Objectives: Evaluate the effects of active-rTMS compared to sham-rTMS among stroke survivors with NOAB, the interventions' cost-effectiveness and explore their experiences qualitatively.

DETAILED DESCRIPTION:
Summary Background: Neurogenic overactive bladder (NOAB) presents with urgency incontinence. Existing NOAB management is expensive, lacks standardized regimens, or is invasive. Therefore, evaluating the effectiveness of non-invasive repetitive transcranial magnetic stimulation (rTMS) for NOAB management among stroke survivors remains crucial.

Objectives: Evaluate the effects of active-rTMS compared to sham-rTMS among stroke survivors with NOAB, the interventions' cost-effectiveness and explore their experiences qualitatively.

Hypothesis: Active-rTMS will reduce NOAB symptom severity for stroke survivors, interventions' cost and assist in gaining insight into the NOAB patients' experiences.

Methods: This study will be a randomised-sham-controlled, double-blinded trial, with embedded qualitative and cost-effectiveness studies. Snowball-convenience sampling technique and computer-generated randomisation will be adopted to recruit 30 participants into active-rTMS and sham-rTMS groups each. Active-rTMS participants will receive a continuous 1 pulse per second 1200 pulses of low-frequency rTMS to the pelvic floor muscle representation in the contralesional primary motor cortex (M1) for 20 minutes thrice weekly. Sham-rTMS participants will receive the same parameters as the active-rTMS group, however, the coil will be rotated 90° away from the scalp. Fifteen active-rTMS participants will be invited for 45-60 minutes focus group discussions. The primary and secondary outcomes will be urinary incontinence severity and quality of life evaluated using the Overactive Bladder Symptom Score and Incontinence-Quality of life Questionnaire, respectively. Quality-adjusted life-years (QALY) will be the cost-effectiveness outcome. The EQ-5D-5L responses will estimate the gain or loss of QALY. A follow-up assessment will be conducted one-months post-intervention. The Client Service Receipt Inventory (CSRI) will be used to collect information on the whole range of services and support required by the study participants.

Statistical analysis: Normality will be evaluated using Shapiro-Wilk test. To determine active-rTMS and sham-rTMS group differences, between-groups analysis of covariance (ANCOVA) will be conducted using R software. Bonferroni correction will be applied for multiple comparisons. Thematic analysis will be used for analysing the qualitative data. For the cost-effectiveness analysis, the unadjusted mean costs and cost differences between active-rTMS and the sham-rTMS group will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors aged between 18-80 years diagnosed with NOAB
* Urodynamic findings confirming detrusor overactivity
* Experience moderate (OABSS scores: 6-11 points) to severe NOAB (OABSS scores: 12 points and above)
* Obtain a Mini-Mental State Examination (MMSE) score of ≥ 24
* Be willing to be randomized

Exclusion Criteria:

* Presence of metals in the cranium, intracardiac lines, increased intracranial pressure, heart diseases, or cardiac pacemaker, use of sacral neuro-modulation
* Pregnancy or less than six months postpartum stage
* Patients with a family history of epilepsy or seizures
* Patients taking tricyclic antidepressants or neuroepileptics
* Participation in any other research project related to urinary incontinence; contra-indicated to MRI, urologic cancer, prostatic pathology, severe pelvic pain, six weeks post-surgery and non-neurogenic bladder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Overactive bladder symptom score (OABSS) questionnaire. | Pre intervention, post intervention (4 weeks) and follow up (4 weeks)
  The OABSS is reported to be a reliable and valid questionnaire for the quantitative evaluation of overactive bladder symptoms in the Hong Kong population (ICC score: 0.82). The measure comprised four questions on OAB symptoms with domain maximum scores ranging from 2 to 5: daytime frequency (two points), night-time frequency (three points), urgency (five points), and UUI (five points). The OABSS total score ranges from 0 to 15 points, with higher scores indicating higher symptom severity. According to severity, mild is defined as a score of 3 to 5 points, moderate as a score of 6 to 11 points, and severe as a score of 12 or more points.

SECONDARY OUTCOMES:
Incontinence Quality-of-Life Questionnaire (I-QoL) | Pre intervention, post intervention (4 weeks) and follow up (4 weeks)
  The I-QoL is reported to be a psychometrically robust incontinence-specific outcome measure for the evaluation of OAB quality of life. The I-QoL measure has 22 items subdivided into 3 subscale scores. The total scores is 100 with 0 representing worst quality of life and 100 means absence of problem (intraclass correlation coefficient [ICC] = 0.93). The measure is tested among Chinese population and found to be of sound psychometric properties; high internal consistency (Cronbach's α: 0.963; excellent test-retest reliability (ICC: 0.74-0.96, P<0.01) and acceptable construct validity.
The Brief Resilience Scale | Pre intervention, post intervention (4 weeks) and follow up (4 weeks)
  The Brief Resilience Scale has been reported to provide unique and critical information regarding "people coping with health-related stressors". Items 1, 3, and 5 on the scale are positively worded. In contrast, items 2, 4, and 6 are negatively worded. Resilience represents coping strategy of individuals to stressed environment and negative life events. The resilience is observed to be lacking in people with urinary incontinence of all age groups
The 5-level EQ-5D (EQ-5D-5L) | Pre intervention, post intervention (4 weeks) and follow up (4 weeks)
  The 5-level EQ-5D (EQ-5D-5L) version developed by the EuroQol Research Foundation will be used to estimate the Quality-adjusted life-years (QALY) gain or loss.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Przydacz M, Denys P, Corcos J. What do we know about neurogenic bladder prevalence and management in developing countries and emerging regions of the world? Ann Phys Rehabil Med. 2017 Sep;60(5):341-346. doi: 10.1016/j.rehab.2017.02.008. Epub 2017 Jun 13. PMID 28623162
- [Background] Brittain KR, Perry SI, Peet SM, Shaw C, Dallosso H, Assassa RP, Williams K, Jagger C, Potter JF, Castleden CM. Prevalence and impact of urinary symptoms among community-dwelling stroke survivors. Stroke. 2000 Apr;31(4):886-91. doi: 10.1161/01.str.31.4.886. PMID 10753993
- [Background] Manack A, Motsko SP, Haag-Molkenteller C, Dmochowski RR, Goehring EL Jr, Nguyen-Khoa BA, Jones JK. Epidemiology and healthcare utilization of neurogenic bladder patients in a US claims database. Neurourol Urodyn. 2011 Mar;30(3):395-401. doi: 10.1002/nau.21003. Epub 2010 Sep 29. PMID 20882676
- [Background] Takahashi S, Kitamura T. Overactive bladder: magnetic versus electrical stimulation. Curr Opin Obstet Gynecol. 2003 Oct;15(5):429-33. doi: 10.1097/00001703-200310000-00012. PMID 14501247
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Nardone R, Versace V, Sebastianelli L, Brigo F, Golaszewski S, Christova M, Saltuari L, Trinka E. Transcranial magnetic stimulation and bladder function: A systematic review. Clin Neurophysiol. 2019 Nov;130(11):2032-2037. doi: 10.1016/j.clinph.2019.08.020. Epub 2019 Sep 3. PMID 31541980
- [Background] Klomjai W, Katz R, Lackmy-Vallee A. Basic principles of transcranial magnetic stimulation (TMS) and repetitive TMS (rTMS). Ann Phys Rehabil Med. 2015 Sep;58(4):208-213. doi: 10.1016/j.rehab.2015.05.005. Epub 2015 Aug 28. PMID 26319963
- [Background] Yani MS, Wondolowski JH, Eckel SP, Kulig K, Fisher BE, Gordon JE, Kutch JJ. Distributed representation of pelvic floor muscles in human motor cortex. Sci Rep. 2018 May 8;8(1):7213. doi: 10.1038/s41598-018-25705-0. PMID 29740105
- [Background] Griffiths D. Neural control of micturition in humans: a working model. Nat Rev Urol. 2015 Dec;12(12):695-705. doi: 10.1038/nrurol.2015.266. Epub 2015 Dec 1. PMID 26620610
- [Background] Griffiths D, Clarkson B, Tadic SD, Resnick NM. Brain Mechanisms Underlying Urge Incontinence and its Response to Pelvic Floor Muscle Training. J Urol. 2015 Sep;194(3):708-15. doi: 10.1016/j.juro.2015.03.102. Epub 2015 Mar 28. PMID 25828973
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Kannan P, Cheung KK, Lau BW, Li L, Chen H, Sun F. A mixed-methods study to evaluate the effectiveness and cost-effectiveness of aerobic exercise for primary dysmenorrhea: A study protocol. PLoS One. 2021 Aug 16;16(8):e0256263. doi: 10.1371/journal.pone.0256263. eCollection 2021. PMID 34398930
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Yani MS, Fenske SJ, Rodriguez LV, Kutch JJ. Motor cortical neuromodulation of pelvic floor muscle tone: Potential implications for the treatment of urologic conditions. Neurourol Urodyn. 2019 Aug;38(6):1517-1523. doi: 10.1002/nau.24014. Epub 2019 May 1. PMID 31044482
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A. Screening questionnaire before TMS: an update. Clin Neurophysiol. 2011 Aug;122(8):1686. doi: 10.1016/j.clinph.2010.12.037. Epub 2011 Jan 11. No abstract available. PMID 21227747
- [Background] Xu L, Fu C, Zhang Q, Xiong F, Peng L, Liang Z, Chen L, He C, Wei Q. Efficacy of biofeedback, repetitive transcranial magnetic stimulation and pelvic floor muscle training for female neurogenic bladder dysfunction after spinal cord injury: a study protocol for a randomised controlled trial. BMJ Open. 2020 Aug 5;10(8):e034582. doi: 10.1136/bmjopen-2019-034582. PMID 32759239